CLINICAL TRIAL: NCT05713045
Title: Late Vitamin K Deficiency-related Bleeding in Neonates (VKDB): Comparison of Four Different Strategies to Prophylaxis Measuring Proteins Induced by Vitamin K Absence (PIVKA)
Brief Title: Late Vitamin K Deficiency-related Bleeding in Neonates (VKLB): Comparison of Different Strategies to Prophylaxis
Acronym: VKLB
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Serafina Perrone, Director of Neonatology Unity, Department of Medicine and Surgery, University of Parma, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: 12150
Record Dates: First submitted 2023-01-24; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Late Vitamin K Deficiency-related Bleeding
MeSH Terms: interventions — Vitamin K 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- intramuscolar injection: intramuscolar injection of 1 mg vitamin K at birth
  Interventions: Dietary Supplement: Konakion
- intramuscolar injection following by oral low dose: intramuscolar injection of 1 mg vitamin K at birth followed by 50 μg/die orally from the second to the fourteenth week of life
  Interventions: Dietary Supplement: Konakion
- intramuscolar injection following by oral high dose: intramuscolar injection of 1 mg vitamin K at birth followed by 150 μg/die orally from the second to the fourteenth week of life
  Interventions: Dietary Supplement: Konakion
- oral administration: oral dose of 2 mg vitamin K at birth, followed by a second dose at 4 weeks, and a third dose at 12 weeks
  Interventions: Dietary Supplement: Konakion

INTERVENTIONS:
Dietary Supplement: Konakion — Comparing 4 different regimen of Vitamin K administration in newborn

SUMMARY:
The goal of this multicentric observational study was to compare four vitamin K dosing regimens in exclusively breastfed healthy term newborns. The main questions it aims to answer were:

* comparing protein induced by vitamin K absence (PIVKA) levels in the different prophylaxis protocols at 48 hours, 1 month and 4 months
* to investigate the compliance and safety of oral vitamin K 1 administration Participants received vitamin K prophilaxis according to birth Hospital regimen. A blood sample was taken at 48 hours, 1 month and 3 months of life. Plasmatic PIVKA-II concentretion was be dosed

Researchers compared four groups of Vitamin K dosing regimens:

1. an intramuscolar injection of 1 mg vitamin K at birth
2. an intramuscolar injection of 1 mg vitamin K at birth followed by 50 μg/die orally from the second to the fourteenth week of life.
3. an intramuscolar injection of 1 mg vitamin K at birth followed by 150 μg/die orally from the second to the fourteenth week of life.
4. an oral dose of 2 mg vitamin K at birth, followed by a second dose at 4 weeks, and a third dose at 12 weeks to see if there is PIVKA-II plasmatic concentration differences.

DETAILED DESCRIPTION:
Partecipanting Centers

* Azienda Ospedaliera Universitaria di Parma
* Azienda Ospedaliera Universitaria di Siena
* Ospedale Buon Consiglio Fatebenefratelli, Napoli
* Ospedale Di Venere, Bari

Materials and Methods Term healthy newborn born from March 2019 to June 2021 was enrolled Vitamin K formulation was Konakion 2 mg/0,2 ml MM paediatric, solution for injection or oral administration, Cheplapharm Arzneimittel GMBH

PIVKA level was was measured on blood drops obtained by heel prick at 48 hours of life, 1 month and 3 months, using the PIVKA-II ELISA Kit, MyBiosource, San Diego, CA, USA.

Blood samples (0,5 ml) were collected in Lithium Heparine draw. After centrifugation at 1000 rpm for 15 minutes plasma was frozen and stored at -20°C. The samples were subsequently analyzed in the Laboratorio di Patologia Clinica, Università degli Studi di Siena.

Medication adherence was measured by questionnaires administrated to parents at 1 month and 3 months of life. A protocol violation (lack of vitamin K administration, concomitant use of other drugs except vitamins, ormula milk or mixed milk feeding) led to exclution of patients

Addictional collected data were:

* sex
* gestational age
* mode of delivery
* Apgar score
* antenatal corticosteroids
* antenatal antibiotics or others drugs
* birth weight
* premature rupture of membranes

Statistical analysis:

Statistical analysis was performed using SPSS 23.0 (IBM, Chicago, IL, USA) and MATLAB 8.0 (The MathWorks, Inc., Natick, MA, USA).

Data were tested for normality with the Shapiro-Wilk test, with the results expressed as mean and standard deviation, median and interquartile range, or frequency and percentage. Data were analyzed using Student's t-test or Wilcoxon rank-sum test for continuous data, and chi-square or Fisher's exact test for categorical variables. A two-tailed p-value <0.05 was considered significant. PIVKA levels were analyzed with repeated measures-ANOVA: different administration regimen was inserted as covariate.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 37+ 0/7 and 42+ 0/7 weeks
* exclusive breastfeeding
* Informed consent by at least one parent

Exclusion Criteria:

* gestational age less than 37+ 0/7 weeks or more than 42+0/7 weeks
* neonatal disease
* liver disease
* formula milk or mixed milk feeding
* withdrawal of informed consent

Ages: 1 Day to 1 Day | Sex: All
Age Groups: Child
Study Population: Term healthy newborn born from March 2019 to June 2021
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
comparing protein induced by vitamin K absence (PIVKA) levels in the different prophylaxis protocols at 48 hours, 1 month and 4 months | 48 hours of life
  PIVKA-II level measured by blood samples
comparing protein induced by vitamin K absence (PIVKA) levels in the different prophylaxis protocols at 48 hours, 1 month and 4 months | 1 month of life
  PIVKA-II level measured by blood samples
comparing protein induced by vitamin K absence (PIVKA) levels in the different prophylaxis protocols at 48 hours, 1 month and 4 months | 3 months of life
  PIVKA-II level measured by blood samples

SECONDARY OUTCOMES:
to investigate the compliance and safety of oral vitamin K 1 administration | 48 hours of life
  Medication Adherence Questionnaire
to investigate the compliance and safety of oral vitamin K 1 administration | 1 month of life, 3 month of life
  Medication Adherence Questionnaire
to investigate the compliance and safety of oral vitamin K 1 administration | 3 months of life
  Medication Adherence Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Pr Serafina Perrone, Parma, Italy

REFERENCES:
- [Background] Lembo C, Buonocore G, Perrone S. The challenge to define the optimal prophylactic regimen for vitamin K deficiency bleeding in infants. Acta Paediatr. 2021 Apr;110(4):1113-1118. doi: 10.1111/apa.15566. Epub 2020 Oct 6. PMID 32892390
- [Background] Shearer MJ. Vitamin K deficiency bleeding (VKDB) in early infancy. Blood Rev. 2009 Mar;23(2):49-59. doi: 10.1016/j.blre.2008.06.001. Epub 2008 Sep 19. PMID 18804903
- [Background] American Academy of Pediatrics Committee on Fetus and Newborn. Controversies concerning vitamin K and the newborn. American Academy of Pediatrics Committee on Fetus and Newborn. Pediatrics. 2003 Jul;112(1 Pt 1):191-2. PMID 12837888
- [Background] Mihatsch WA, Braegger C, Bronsky J, Campoy C, Domellof M, Fewtrell M, Mis NF, Hojsak I, Hulst J, Indrio F, Lapillonne A, Mlgaard C, Embleton N, van Goudoever J; ESPGHAN Committee on Nutrition. Prevention of Vitamin K Deficiency Bleeding in Newborn Infants: A Position Paper by the ESPGHAN Committee on Nutrition. J Pediatr Gastroenterol Nutr. 2016 Jul;63(1):123-9. doi: 10.1097/MPG.0000000000001232. PMID 27050049